CLINICAL TRIAL: NCT04233775
Title: Altered Cerebral Growth and Development in Infants With Congenital Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Walter Knirsch, Professor, University Children's Hospital, Zurich
Other Study IDs: Knirsch 01
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Neurodevelopmental Disorders; Congenital Heart Disease; Brain Injuries; Fetal Growth Retardation
Keywords: congenital heart disease; brain imaging; neurodevelopmental outcome
MeSH Terms: conditions — Neurodevelopmental Disorders; Heart Defects, Congenital; Brain Injuries; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Congenital heart disease (CHD) is the most frequent inborn defect with an incidence of 1 in 100 newborns per year, i.e. 800 children born in Switzerland per year. 10% to 15% of cases are born with single ventricle (SV), the most complex type of CHF requiring immediate surgical intervention after birth. Infants with SV CHD are treated in three surgical staged procedures over the first three years of life. However, cerebral injuries occur in around 40% of those children and impact neurocognitive abilities. As more than 90% of all infants with CHD survive to adulthood, scientific concern is focussed on patient-individual course brain growth and development within the relative contribution of fetal, perinatal, cardiac and surgical risk factors. Therefore, serial cerebral MRI examinations are needed, starting (1) at the third trimester during fetal life proceeding to (2) pre- and postoperative time points at the stage I surgery after birth and (3) before stage II surgery at 4 months of age. We will compare the cerebral MRI findings with a healthy control population, recruited at the same time points, and correlate brain growth and development with the neurodevelopmental outcome assessed at one year of age. Three Pediatric Heart Centers in Switzerland and Germany will participate.

The overall aims are:

1. To analyse the patient-individual cerebral developmental trajectories, brain growth and determine the time course of brain abnormalities in infants with single ventricle CHD by serial cerebral MRI during fetal life, after birth and at an age of 4 months (primary endpoints).
2. To determine the neurodevelopmental outcome at one year of age using the Bayley III and will be correlated with the brain growth and brain development in the third trimester of fetal life and at the age of 4 months (secondary endpoints).
3. To analyse fetal, neonatal, surgery-related and intensive care associated factors determining the patient-individual course for altered cerebral growth and impaired neurodevelopmental outcome at one year of age.

Methodology: We will prospectively enroll fetuses and neonates with single ventricle CHD at the three Pediatric Heart Centers in Switzerland (Zurich, Bern) and Germany (Giessen). Advanced MR imaging will assess cerebral volumes, microstructural and hemodynamic changes at repeated time points during the third trimester of fetal life (32. week of gestation), the perioperative neonatal period before and after stage I surgery and before stage II surgery at 4 months of age. Biomechanical analysis of longitudinal changes of brain morphology will be applied to longitudinal fetal and neonatal MRI data. Outcome is determined with the Bayley-III at one year of age.

Significance: Using a population-based sample of children with single ventricle CHD, we will be able to determine cerebral growth from the third fetal trimester until the first 4 months after birth, when the brain is most rapidly growing. By performing serial brain imaging, the knowledge of etiological pattern affecting cerebral growth, development and brain injury will increase. Morphometric and biomechanical analysis of brain growth patterns will be performed that may capture fine-grained changes associated with CHD. By correlating these data with the neurodevelopmental outcome at one year of age it will be possible to identify specific risk constellations leading to impaired brain development and categories of brain injuries that confer a higher risk of adverse outcome. The better understanding of the pathophysiological mechanisms will serve as the basis for neuroprotective studies and pharmacological trials aiming to improve outcomes in children with CHD in the future.

ELIGIBILITY:
Inclusion Criteria:

All fetuses and neonates with the diagnosis complex type of CHD undergoing open-heart surgery are prospectively enrolled

Exclusion Criteria:

a) Clinical evidence or suspicion of a congenital malformation or syndrome, b) brain malformation, c) congenital infection and d) preterms before 37 weeks. These criteria will exclude fetuses and newborns with other conditions that will impact neurodevelopmental outcome.

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fetuses and neonates with complex type of CHD form the study population group. Healthy control population will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-individual cerebral developmental trajectories | 6 months
  Brain growth and brain development from third trimester of fetal life to 4 months after birth will be analysed

SECONDARY OUTCOMES:
Neurodevelopmental outcome at one year of age using the Bayley III | One year
  Bayley Scales Bayley scales of Infant Development will be used as a standardized method to assess cognitive and motor development in infants.
Risk factor analysis | One year
  Risk factor analysis of fetal, neonatal, surgery-related and intensive care associated factors determining the patient-individual course for altered cerebral growth and impaired neurodevelopmental outcome at one year of age

CONTACTS AND LOCATIONS:
Overall Officials: Walter H Knirsch, MD, Principal Investigator — University Children's Hospital, Pediatric Heart Center, Pediatric Cardiology
Locations (1):
- University Children's Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knirsch W, De Silvestro A, Steger C, Rathke V, Weber R, Von Rhein M, Schneider J, Hutter D, Reich B, Held U, Hackenberg A, Tuura O'Gorman R, Kottke R, Jakab A; BrainCHD Study Group. Serial cerebral magnetic resonance imaging before and after birth in patients with complex congenital heart disease - a prospective, multicentre observational study. Swiss Med Wkly. 2025 Dec 2;155:4466. doi: 10.57187/s.4466. PMID 41397378